CLINICAL TRIAL: NCT01647516
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo Controlled Parallel-Group Study to Evaluate the Clinical Efficacy and Safety of Induction Therapy With RPC1063 in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: Efficacy and Safety Study of Ozanimod in Ulcerative Colitis
Acronym: Touchstone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPC01-202
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ozanimod 0.5 mg (Experimental): Participants received 0.5 mg capsules of ozanimod hydrochloride daily during the induction period weeks 0-9 (an initial 8-day dose escalation regimen in the induction period that consisted of 4 days of ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg), followed by 3 days of ozanimod HCl 0.5 mg, (equivalent to ozanimod 0.46 mg) followed by the assigned treatment level for at least 8 weeks. Participants who completed the induction period and were responders at week 8, continued to receive the same dose of ozanimod during the maintenance period up to week 32. Participants who received ozanimod 0.5 mg capsules and completed the induction period and were non-responders at Week 8 and who completed the maintenance period or experienced a disease relapse, were given the option to enter the OLP and receive 1 mg ozaninod capsules daily up to 6 years. Participants who had not shown clinical improvement 8 weeks after initiation of the OLP were discontinued from the study.
  Interventions: Drug: Ozanimod
- Ozanimod 1 mg (Experimental): Participants received 1 mg capsules of ozanimod hydrochloride daily during the induction period weeks 0-9 (an initial 8-day dose escalation regimen in the induction period that consisted of 4 days of ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg), followed by 3 days of ozanimod HCl 0.5 mg, (equivalent to ozanimod 0.46 mg) followed by the assigned treatment level for at least 8 weeks. Participants who completed the induction period and were responders at week 8, continued to receive the same dose of ozanimod during the maintenance period up to week 32. Participants who received ozanimod 1 mg capsules and completed the induction period and were non-responders at Week 8 and who completed the maintenance period or experienced a disease relapse, were given the option to enter the OLP and receive 1 mg ozaninod capsules daily up to 6 years. Participants who had not shown clinical improvement 8 weeks after initiation of the OLP were discontinued from the study.
  Interventions: Drug: Ozanimod
- Placebo (Placebo Comparator): Identically matching placebo capsules daily for 32 weeks followed by an optional open label treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ozanimod — Ozanimod capsules by mouth daily.
  Other Names: Zeposia, RPC 1063
  Arms: Ozanimod 0.5 mg; Ozanimod 1 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether RPC1063 is effective in the treatment of ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis (UC) confirmed on endoscopy
* Moderately to severely active UC (Mayo score 6-12)

Exclusion Criteria:

* Current use of anti-TNF agents

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2012-12-26 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AnnKatrin Petersen, MD, Study Director — Bristol-Myers Squibb
Locations (88):
- United States (10):
  - Anaheim Clinical Trials, Anaheim, California
  - University of California San Diego, La Jolla, California
  - Alliance Clinical Research, Oceanside, California
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Endoscopic Microsurgery Associates, Towson, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Long Island Clinical Research Associates, Great Neck, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
- The Alfred Hospital, Melbourne, Victoria, Australia
- Universitair Ziekenhuis Leuven, Campus Gasthuisberg, Leuven, Belgium
- Bulgaria (9):
  - Multiprofile Hospital for Active Treatment Kaspela, Plovdiv
  - University Multiprofile Hospital for Active Treatment ACIBADEM City Clinic Sofia, Sofia
  - UMHAT Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna ISUL EAD, Sofia
  - Military Medical Academy, Sofia
  - Multiprofile Hospital for Active Treatment Doverie AD, Sofia
  - Multiprofile Hospital for Active Treatment Sveti Panteleimon - Sofia AD, Sofia
  - Multiprofile Hospital for Active Treatment Sofiamed, Sofia
  - Multiprofile Hospital for Active Treatment Sveta Marina EAD, Varna
- London Health Sciences Centre, University Hospital, London, Ontario, Canada
- Greece (3):
  - Evaggelismos General Hospital, Athens
  - University Hospital of Ioannina, Ioannina
  - University Hospital of Larissa, Larissa
- Hungary (4):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Vasútegészségügyi Nonprofit Kiemelten Közhasznú Kft. Debreceni Egészségügyi Központja, Debrecen
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Ikazia Ziekenhuis, Rotterdam
- New Zealand (5):
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Hutt Valley District Health Board, Lower Hutt
  - North Shore Hospital, Milford
- Poland (12):
  - SPZOZ Wojewodzki Szpital Zespolony im. J.Sniadeckiego, Bialystok
  - Niepubliczny Zaklad Opieki Zdrowotnej INTERMED, Częstochowa
  - Elblaski Szpital Specjalistyczny z Przychodnia, Elblag
  - Przychodnia Lekarska Nowy Chelm, Gdansk
  - Economicus - NZOZ ALL-MEDICUS, Katowice
  - Centrum Opieki Zdrowotnej Orkan Med, Ksawerów
  - Niepubliczny Zaklad Opieki Zdrowotnej CENTRUM MEDYCZNE Szpital Swietej Rodziny, Lodz
  - Instytut Medycyny Wsi, Lublin
  - MEDICOR Centrum Medyczne, Rzeszów
  - Niepubliczny Zaklad Opieki Zdrowotnej Triclinium, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej VIVAMED, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
- Russia (9):
  - Regional Clinical Hospital, Krasnoyarsk
  - SBEI HPE First Moscow State Medical University n.a. I.M. Sechenov of the MoH of the RF, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. N.A. Semashko, Nizhny Novgorod
  - Novosibirsk State Medical University, Novosibirsk
  - SBEI of HPE Omsk State Medical Academy Ministry of healthcare of RF, Omsk
  - SEIHPE Rostov State Medical University of MoH of RF, Rostov-on-Don
  - Russian Medical Military Academy na SMKirov, Saint Petersburg
  - City Hospital 26, Saint Petersburg
  - Medical Company Hepatolog, Samara
- Slovakia (3):
  - Slovak Research Center, Ilava
  - Specializovana Nemocnica Svorada Zobor, Nitra
  - GASTRO I., s.r.o., Prešov
- South Korea (9):
  - Yeungnam University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Kyunghee University Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - The Catholic University of Korea, St.Vicent's Hospital, Suwon
  - Wonju Christian Hospital, Wŏnju
- Ukraine (12):
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Ivano-Frankivsk City Clinical Hospital #1 Dep of Surgery SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - Institute of Therapy n.a. L.T. Maloy of NAMS of Ukraine, Kharkiv
  - Kyiv CCH #8 Dept of Gastroenterology P.L. Shupyk NMA of PGE, Kyiv
  - Order of the Red Star MMMCC MMCH Clinic of Gastroenterology, Kyiv
  - CNI Consultative and Diagnostic Center of Desnianskyi District of Kyiv, Kyiv
  - Lviv Regional Clinical Hospital, Lviv
  - Communal City Clinical Hospital of Ambulance, Dept of Therapy #1 D.Halytskyi Lviv NMU, Lviv
  - Vinnytsia Regional Clinical, Vinnytsia
  - Medical Clinical Research Center "Health Clinic", Vinnytsia
  - Municipal Institution Zaporizhzhia, Zaporizhzhia
  - Zaporizhzhya city multidisciplinary clinical hospital #9, Zaporizhzhya

REFERENCES:
- [Background] Sandborn WJ, Feagan BG, Wolf DC, D'Haens G, Vermeire S, Hanauer SB, Ghosh S, Smith H, Cravets M, Frohna PA, Aranda R, Gujrathi S, Olson A; TOUCHSTONE Study Group. Ozanimod Induction and Maintenance Treatment for Ulcerative Colitis. N Engl J Med. 2016 May 5;374(18):1754-62. doi: 10.1056/NEJMoa1513248. PMID 27144850
- [Derived] Regueiro M, Siegmund B, Horst S, Moslin R, Charles L, Petersen A, Tatosian D, Wu H, Lawlor G, Fischer M, D'Haens G, Colombel JF. Concomitant Administration of Ozanimod and Serotonergic Antidepressants in Patients With Ulcerative Colitis or Relapsing Multiple Sclerosis. Inflamm Bowel Dis. 2025 Apr 10;31(4):1010-1017. doi: 10.1093/ibd/izae136. PMID 39018016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 57 sites from 13 countries located in Europe, North America, and the Asia-Pacific region.
Pre-assignment Details: Participants were randomly assigned in a 1:1:1 ratio on Day 1 to placebo, ozanimod 0.5 mg, or ozanimod 1 mg capsules and were stratified by whether they had received anti-tumor necrosis factor class of therapy (yes vs no).
Groups:
- Placebo: Participants received identically matching placebo capsules daily for 9 weeks during the induction period (weeks 0 to 9). Participants who completed the induction period and were responders, continued to receive identically matching placebo tablets during the maintenance period (weeks 9-32).
- Ozanimod Hydrochloride 0.5 mg: Participants received 0.5 mg capsules of ozanimod hydrochloride daily during the induction period weeks 0-9 (an initial 8-day dose escalation regimen in the induction period that consisted of 4 days of ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg), followed by 3 days of ozanimod HCl 0.5 mg, (equivalent to ozanimod 0.46 mg) followed by the assigned treatment level for at least 8 weeks. Participants who completed the induction period and were responders at week 8, continued to receive the same dose of ozanimod during the maintenance period up to week 32.
- Ozanimod Hydrochloride 1 mg: Participants received 1 mg capsules of ozanimod hydrochloride daily during the induction period weeks 0-9 (an initial 8-day dose escalation regimen in the induction period that consisted of 4 days of ozanimod HCl 0.25 mg (equivalent to ozanimod 0.23 mg), followed by 3 days of ozanimod HCl 0.5 mg, (equivalent to ozanimod 0.46 mg) followed by the assigned treatment level for at least 8 weeks. Participants who completed the induction period and were responders at week 8, continued to receive the same dose of ozanimod during the maintenance period up to week 32.
- Open-Label Treatment Period (OLP): Placebo/Ozanimod: Participants who received placebo capsules and completed the induction period and were non-responders at week 8 and those who completed the maintenance period or experienced a disease relapse, were given the option to enter the open label treatment period (OLP) and receive 1 mg ozanimod daily up to 6 years. Participants who had not shown clinical improvement 8 weeks after initiation of the OLP were discontinued from the study.
- OLP: Ozanimod 0.5 mg/Ozanimod 1 mg: Participants who received ozanimod 0.5 mg capsules and completed the induction period and were non-responders at week 8 and who completed the maintenance period or experienced a disease relapse, were given the option to enter the OLP and receive 1 mg ozaninod capsules daily up to 6 years. Participants who had not shown clinical improvement 8 weeks after initiation of the OLP were discontinued from the study.
- OLP: Ozanimod 1 mg/Ozanimod 1 mg: Participants who received 1 mg ozanimod capsules and completed the induction period and were non-responders at week 8 and those who completed the maintenance period or experienced a disease relapse, were given the option to enter the open label treatment period (OLP) and continue to receive 1 mg ozaninod daily up to 6 years. Participants who had not shown clinical improvement 8 weeks after initiation of the OLP were discontinued from the study.
Period: Induction Period (IP)
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg | Open-Label Treatment Period (OLP): Placebo/Ozanimod | OLP: Ozanimod 0.5 mg/Ozanimod 1 mg | OLP: Ozanimod 1 mg/Ozanimod 1 mg
Started | 66 | 66 | 67 | 0 | 0 | 0
Received Study Drug | 65 | 65 | 67 | 0 | 0 | 0
Completed | 60 | 63 | 63 | 0 | 0 | 0
Not Completed | 6 | 3 | 4 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 3 | 0 | 0 | 0
Not completed — Participant Choice | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — No study drug received | 1 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Period (MP)
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg | Open-Label Treatment Period (OLP): Placebo/Ozanimod | OLP: Ozanimod 0.5 mg/Ozanimod 1 mg | OLP: Ozanimod 1 mg/Ozanimod 1 mg
Started | 25 (The MP includes participants who were responders at week 8.) | 36 (The MP includes participants who were responders at week 8.) | 42 (The MP includes participants who were responders at week 8.) | 0 | 0 | 0
Completed | 21 | 30 | 40 | 0 | 0 | 0
Not Completed | 4 | 6 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 4 | 1 | 0 | 0 | 0
Period: Open-Label Period
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg | Open-Label Treatment Period (OLP): Placebo/Ozanimod | OLP: Ozanimod 0.5 mg/Ozanimod 1 mg | OLP: Ozanimod 1 mg/Ozanimod 1 mg
Started | 0 | 0 | 0 | 55 (The participants were: non-responders at Week 8,completed the MP or had disease relapse during MP) | 56 (The participants were: non-responders at Week 8,completed the MP or had disease relapse during MP) | 59 (The participants were: non-responders at Week 8,completed the MP or had disease relapse during MP)
Completed | 0 | 0 | 0 | 6 | 5 | 3
Not Completed | 0 | 0 | 0 | 49 | 51 | 56
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 6 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 9 | 11 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Sponsor Termination; moved to 3102 study | 0 | 0 | 0 | 18 | 13 | 23
Not completed — Lack of Efficacy | 0 | 0 | 0 | 7 | 9 | 10
Not completed — Participant Choice to Stop Study Drug | 0 | 0 | 0 | 7 | 9 | 10
Not completed — No completion / discontinuation visit | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat ( ITT) population consisted of all randomized patients who received at least one dose of study treatment, with treatment assignment designated according to randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg | Total
Number analyzed (Participants) | 65 | 65 | 67 | 197
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.9 (12.30) | 38.8 (12.06) | 41.8 (11.01) | 40.8 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 33 | 19 | 82
  Male | 35 | 32 | 48 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 63 | 64 | 67 | 194
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61 | 59 | 62 | 182
  Black | 2 | 1 | 1 | 4
  Asian | 2 | 3 | 3 | 8
  Other | 0 | 1 | 1 | 2
  Missing | 0 | 1 | 0 | 1
Years Since Ulcerative Colitis Diagnosis [Mean (Standard Deviation); unit: Years] | 6.1 (5.46) | 5.9 (5.44) | 6.7 (6.76) | 6.2 (5.91)
Any Prior Ulcerative Colitis Medication Use [Count of Participants; unit: Participants]
  Aminosalycylates | 63 | 63 | 67 | 193
  Systemic Corticosteroids | 52 | 49 | 52 | 153
  Azathioprine | 17 | 23 | 19 | 59
  Anti-Tumor Necrosis Factors (Anti-TNF) | 10 | 12 | 15 | 37
  6-Mercaptopurine | 2 | 1 | 5 | 8
  Other Immunomodulators | 6 | 5 | 3 | 14
  Topical Medication | 3 | 0 | 0 | 3
  Methotrexate | 1 | 1 | 0 | 2
Mayo Score [Mean (Standard Deviation); unit: Units on a Scale] — The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  Units on a Scale | 8.6 (1.51) | 8.3 (1.45) | 8.5 (1.61) | 8.5 (1.52)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission Based on the Central Read of the Mayo Score (MS), at Week 8
Description: Clinical Remission was defined as: Mayo score of <2 points and with no individual subscore of > 1 point.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  * Stool Frequency Subscore (SFS)
  * Rectal bleeding Subscore (RBS)
  * Endoscopy Subscore
  * Physician's Global Assessment (PGA)
  Clinical Remission was based on the 4-component Mayo definition.
Time Frame: Week 8
Population: The intent to treat ( ITT) population consisted of all randomized participants who received at least one dose of study treatment, with treatment. Participants with missing Mayo scores were classified as non-responders.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 65 | 65 | 67
Percentage of Participants | 6.2 | 13.8 | 16.4
Statistical Analysis 1: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority; p = 0.0482, Cochran-Mantel-Haenszel; Stratified by prior anti-tumor necrosing factor (anti-TNF) therapy experience, (yes or no); Odds Ratio (OR) = 3.262, 95% CI 2-sided [0.969 to 10.984]
Statistical Analysis 2: Comparison: Placebo vs Ozanimod Hydrochloride 0.5 mg; Test type: Superiority; p = 0.1422, Cochran-Mantel-Haenszel; Stratified by prior anti-tumor necrosing factor (anti-TNF) therapy experience, (yes or no); Odds Ratio (OR) = 2.500, 95% CI 2-sided [0.722 to 8.661]

2. Secondary Outcome: Percentage of Participants Who Achieved a Clinical Response in the Mayo Score (MS) at Week 8
Description: Clinical response was defined as a reduction from baseline in Mayo score ≥3 points and ≥30%, and a decrease from baseline in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of ≤ 1 point.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  Clinical Respone was based on the 4-component Mayo definition.
Time Frame: Week 8
Population: The ITT population consisted of all randomized participants who received at least one dose of study treatment, with treatment assignment designated according to randomized treatment. Participants with missing Mayo score were considered non-responders. Non responder imputation (NRI).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 65 | 65 | 67
Percentage of Participants | 36.9 | 53.8 | 56.7
Statistical Analysis 1: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority; p = 0.0207, Cochran-Mantel-Haenszel; Stratified by prior anti-tumor necrosing factor (anti-TNF) therapy experience, (yes or no); Odds Ratio (OR) = 2.158, 95% CI 2-sided [1.093 to 4.263]
Statistical Analysis 2: Comparison: Placebo vs Ozanimod Hydrochloride 0.5 mg; Test type: Superiority; p = 0.0648, Cochran-Mantel-Haenszel; Stratified by prior anti-tumor necrosing factor (anti-TNF) therapy experience, (yes or no); Odds Ratio (OR) = 1.947, 95% CI 2-sided [0.961 to 3.946]

3. Secondary Outcome: Change From Baseline in Mayo Score at Week 8
Description: The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  * Stool Frequency Subscore (SFS)
  * Rectal bleeding Subscore (RBS)
  * Endoscopy Subscore
  * Physician's Global Assessment (PGA)
Time Frame: Baseline to Week 8
Population: The ITT population consisted of all randomized patients who received at least one dose of study treatment, with treatment assignment designated according to randomized treatment. Includes participants with available data.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 62 | 64 | 65
Units on a Scale | -2.0 (2.52) | -2.6 (2.92) | -3.4 (2.79)
Statistical Analysis 1: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority; p = 0.0042, ANCOVA; The analysis of covariance model, adjusting for baseline Mayo score and prior anti-TNF (yes or no)
Statistical Analysis 2: Comparison: Placebo vs Ozanimod Hydrochloride 0.5 mg; Test type: Superiority; p = 0.1415, ANCOVA; The analysis of covariance model, adjusting for baseline Mayo score and prior anti-TNF (yes or no)

4. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 8
Description: Mucosal healing is defined as an endoscopy subscore ≤ 1 point. Endoscopy subscores were calculated based on central endoscopy reading.
  The endoscopy scale:
  0 = Normal or inactive disease
  1. = Mild disease (erythema, decreased vascular pattern, mild friability)
  2. = Moderate disease (marked erythema, lack of vascular pattern, friability, erosions)
  3. = Severe disease (spontaneous bleeding, ulceration)
Time Frame: Week 8
Population: The ITT population consisted of all randomized patients who received at least one dose of study treatment, with treatment assignment designated according to randomized treatment. Non-responder imputation (NRI).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 65 | 65 | 67
Percentage of Participants | 12.3 | 27.7 | 34.3
Statistical Analysis 1: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority; p = 0.0023, Cochran-Mantel-Haenszel; Stratified by prior anti-TNF therapy experience, (yes or no); Odds Ratio (OR) = 3.861, 95% CI 2-sided [1.572 to 9.484]
Statistical Analysis 2: Comparison: Placebo vs Ozanimod Hydrochloride 0.5 mg; Test type: Superiority; p = 0.0348, Cochran-Mantel-Haenszel; Stratified by prior anti-TNF therapy experience, (yes or no); Odds Ratio (OR) = 2.647, 95% CI 2-sided [1.058 to 6.621]

5. Secondary Outcome: Percentage of Participants Who Achieved Clinical Remission in the Mayo Score at Week 32
Description: Clinical Remission was defined as: Mayo score of <2 points and with no individual subscore of > 1 point.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a score of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  * Stool Frequency Subscore (SFS)
  * Rectal bleeding Subscore (RBS)
  * Endoscopy Subscore
  * Physician's Global Assessment (PGA)
Time Frame: Week 32
Population: The ITT population consisted of all randomized patients who received at least one dose of study treatment, with treatment assignment designated according to randomized treatment. Participants with missing Mayo score were considered non-responders. Non responder imputation (NRI).
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 65 | 65 | 67
Percentage of Participants | 6.2 | 26.2 | 20.9
Statistical Analysis 1: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority; p = 0.0108, Cochran-Mantel-Haenszel; Stratified by prior anti-TNF therapy experience, (yes or no); Odds Ratio (OR) = 4.332, 95% CI 2-sided [1.323 to 14.186]
Statistical Analysis 2: Comparison: Placebo vs Ozanimod Hydrochloride 0.5 mg; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel; Stratified by prior anti-TNF therapy experience, (yes or no); Odds Ratio (OR) = 5.443, 95% CI 2-sided [1.706 to 17.365]

6. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response at Week 32
Description: Clinical response was defined as a reduction from baseline in Mayo score ≥3 points and ≥30%, and a decrease from baseline in the rectal bleeding subscore of ≥ 1 point or an absolute rectal bleeding subscore of ≤ 1 point.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, rectosigmoidoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
  * Stool Frequency Subscore (SFS)
  * Rectal bleeding Subscore (RBS)
  * Endoscopy Subscore
  * Physician's Global Assessment (PGA)
Time Frame: Week 32
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 65 | 65 | 67
Percentage of Participants | 20.0 | 35.4 | 50.7
Statistical Analysis 1: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority — Stratified by prior anti-TNF therapy experience, (yes or no); p = 0.0002, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.030, 95% CI 2-sided [1.871 to 8.678]
Statistical Analysis 2: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority; p = 0.0571, Cochran-Mantel-Haenszel; Stratified by prior anti-TNF therapy experience, (yes or no); Odds Ratio (OR) = 2.154, 95% CI 2-sided [0.974 to 4.763]

7. Secondary Outcome: Percentage of Participants With Mucosal Healing at Week 32
Description: as for outcome 4
Time Frame: Week 32
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 65 | 65 | 67
Percentage of Participants | 12.3 | 32.3 | 32.8
Statistical Analysis 1: Comparison: Placebo vs Ozanimod Hydrochloride 1 mg; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel; Stratified by prior anti-TNF therapy experience, (yes or no); Odds Ratio (OR) = 3.557, 95% CI 2-sided [1.444 to 8.762]
Statistical Analysis 2: Comparison: Placebo vs Ozanimod Hydrochloride 0.5 mg; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel; Stratified by prior anti-TNF therapy experience, (yes or no); Odds Ratio (OR) = 3.428, 95% CI 2-sided [1.384 to 8.494]

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Induction Period
Description: A TEAE was defined as any event with an onset date on or after first dose date or any ongoing event on the first dose date that worsens in severity after first dose date and until 90 days following the last dose of treatment with the study drug. earlier. A serious AE = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs was assessed by the investigator and based on the following scale: Mild = an AE usually transient in nature and generally not interfering with normal activities; Moderate = an AE that is sufficiently discomforting to interfere with normal activities; Severe = an AE that is incapacitating and prevents normal activities.
Time Frame: From the first dose of investigational product (IP) up to 90 days after the last dose of IP or at follow-up visit; the mean total duration of IP exposure was 52.8 days, 56.1 days and 50.8 days respectively for 0.5 mg, 1 mg ozanimod and placebo
Population: Safety population included all participants who were enrolled and received at least 1 dose of investigational product (IP).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 65 | 65 | 67
Participants
  ≥ 1 TEAE | 21 | 24 | 17
  ≥ 1 Moderate or Severe TEAE | 7 | 12 | 6
  ≥ 1 Severe TEAE | 2 | 1 | 1
  ≥ 1 Possibly, Probably or Definitely Related TEAE | 2 | 5 | 5
  ≥ 1 Serious SAE | 4 | 1 | 2
  ≥ 1 Possibly, Probably or Related Serious TEAE | 0 | 0 | 0
  ≥ 1 TEAE Leading to Withdrawal From Study | 1 | 2 | 1
  Death | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAE) During the Maintenance Period
Description: as for outcome 8
Time Frame: From the first dose of IP up to 90 days after the last dose of IP or at follow-up visit; the mean total duration of IP exposure was 156.3 days, 171.1 days and 154.5 days respectively for 0.5 mg, 1 mg ozanimod and placebo.
Population: Safety population included all participants who were enrolled and received at least 1 dose of investigational product (IP) and who entered the maintenance period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ozanimod Hydrochloride 0.5 mg | Ozanimod Hydrochloride 1 mg
Number analyzed (Participants) | 25 | 36 | 42
Participants
  ≥ 1 TEAE | 8 | 4 | 11
  ≥ 1 Moderate or Severe TEAE | 4 | 1 | 5
  ≥ 1 Severe TEAE | 1 | 0 | 1
  ≥ 1 Possibly, Probably or Definitely Related TEAE | 0 | 0 | 2
  ≥ 1 Serious TEAE | 2 | 0 | 1
  ≥ 1 Possibly, Probably or Related Serious TEAE | 0 | 0 | 0
  ≥ 1 TEAE Leading to Withdrawal From Study | 3 | 0 | 0
  Death | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With TEAE During the Open-Label Treatment Period (OLP)
Description: as for outcome 8
Time Frame: From the first dose of IP until 90 days after the last dose of IP or at follow-up visit; the mean total duration of study drug exposure in the OLP was 2.42 years
Population: Safety population included all participants who were enrolled and received at least 1 dose of investigational product (IP). All participants in the OLE safety population received 1 mg capsules ozanimod as noted in the description.
Measure: Count of Participants; unit: Participants
Groups:
- Ozanimod: Participants who completed the induction period and were non-responders at Week 8 and those who completed the maintenance period or experienced a disease relapse entered the open label treatment period (OLP) and received 1 mg ozaninod daily up to 6 years. Participants who did not show clinical improvement 8 weeks after initiation of the OLP were discontinued from the study.
Arm/Group | Ozanimod
Number analyzed (Participants) | 170
Participants
  ≥ 1 TEAE | 101
  ≥ 1 Moderate or Severe TEAE | 63
  ≥ 1 Severe TEAE | 17
  ≥ 1 Possible, Probable or Related TEAE | 27
  ≥ 1 Related TEAE | 2
  ≥ 1 Serious TEAE | 27
  ≥ 1 Related Serious TEAE | 0
  ≥ 1 Possible, Probable or Related Serious TEAE | 4
  ≥ 1 TEAE Leading to Discontinuation of IP | 14
  ≥ 1 TEAE Leading to Withdrawal from Study | 13
  Death | 1
  1 Death Possible, Probable or Related to IP | 1

ADVERSE EVENTS:
Time Frame: From the first dose of investigational product (IP) up to 90 days after the last dose of IP or at follow-up visit; the mean total duration of IP exposure was 52.8 days, 56.1 days and 50.8 days respectively for 0.5 mg, 1 mg ozanimod and placebo during the induction period.
Description: The mean total duration of study drug exposure was 156.3 days, 171.1 days and 154.5 days respectively for 0.5 mg, 1 mg ozanimod and placebo during the maintenance period and 2.42 years during the open label treatment period, The safety population includes all participants who received at least dose of study treatment; maintenance phase data includes all participants who entered the maintenance phase.
Groups:
- Induction Period: Placebo: Participants received identically matching placebo capsules daily for 9 weeks during the induction period (weeks 0 to 9).
- Induction Period: Ozanimod HCL 0.5 mg: Participants received 0.5 mg ozanimod capsules daily during the induction period (weeks 0 to 9).
- Induction Period: Ozanimod HCL 1 mg: Participants received 1 mg ozanimod capsules daily during the induction period (weeks 0 to 9).
- Maintenance Period: Placebo: Participants originally assigned to placebo who completed the induction period and were responders at week 8 continued to receive placebo in the maintenance period. Participants received identically matching placebo capsules daily during the maintenance period (weeks 9-32).
- Maintenance Period: Ozanimod HCL 0.5 mg: Participants originally assigned to ozanimod 0.5 mg who completed the induction period and were responders at week 8 continued to receive ozanimod 0.5 mg daily in the maintenance period. Participants received 0.5 mg ozanimod capsules daily during the maintenance period (weeks 9 to 32).
- Maintenance Period: Ozanimod HCL 1 mg: Participants originally assigned to ozanimod 1 mg who completed the induction period and were responders at week 8 continued to receive ozanimod 0.5 mg daily in the maintenance period. Participants received 1 mg ozanimod capsules daily during the maintenance period (weeks 9 to 32).
- OLP: Ozanimod 1mg/Ozanimod 1 mg: Participants who received 1 mg ozanimod capsules and completed the induction period and were non-responders at Week 8 and those who completed the maintenance period or experienced a disease relapse, were given the option to enter the open label treatment period (OLP) and continue to receive 1 mg ozaninod daily up to 6 years. Participants who had not shown clinical improvement 8 weeks after initiation of the OLP were discontinued from the study.
Arm/Group | Induction Period: Placebo | Induction Period: Ozanimod HCL 0.5 mg | Induction Period: Ozanimod HCL 1 mg | Maintenance Period: Placebo | Maintenance Period: Ozanimod HCL 0.5 mg | Maintenance Period: Ozanimod HCL 1 mg | Open-Label Treatment Period (OLP): Placebo/Ozanimod | OLP: Ozanimod 0.5 mg/Ozanimod 1 mg | OLP: Ozanimod 1mg/Ozanimod 1 mg
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/67 | 0/25 | 0/36 | 0/42 | 0/55 | 1/56 | 0/59
Serious Adverse Events (participants affected / at risk) | 4/65 | 1/65 | 2/67 | 2/25 | 0/36 | 1/42 | 5/55 | 14/56 | 11/59
Other Adverse Events (participants affected / at risk) | 9/65 | 8/65 | 8/67 | 3/25 | 2/36 | 2/42 | 19/55 | 17/56 | 22/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Placebo (N=65) | Induction Period: Ozanimod HCL 0.5 mg (N=65) | Induction Period: Ozanimod HCL 1 mg (N=67) | Maintenance Period: Placebo (N=25) | Maintenance Period: Ozanimod HCL 0.5 mg (N=36) | Maintenance Period: Ozanimod HCL 1 mg (N=42) | Open-Label Treatment Period (OLP): Placebo/Ozanimod (N=55) | OLP: Ozanimod 0.5 mg/Ozanimod 1 mg (N=56) | OLP: Ozanimod 1mg/Ozanimod 1 mg (N=59)
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 3 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Placebo (N=65) | Induction Period: Ozanimod HCL 0.5 mg (N=65) | Induction Period: Ozanimod HCL 1 mg (N=67) | Maintenance Period: Placebo (N=25) | Maintenance Period: Ozanimod HCL 0.5 mg (N=36) | Maintenance Period: Ozanimod HCL 1 mg (N=42) | Open-Label Treatment Period (OLP): Placebo/Ozanimod (N=55) | OLP: Ozanimod 0.5 mg/Ozanimod 1 mg (N=56) | OLP: Ozanimod 1mg/Ozanimod 1 mg (N=59)
Anaemia (Blood and lymphatic system disorders) | 4 | 4 | 1 | 0 | 0 | 0 | 4 | 3 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 3
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 5
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 4
Headache (Nervous system disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 3
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT01647516/Prot_000.pdf
  • Statistical Analysis Plan (2014-09-23): https://cdn.clinicaltrials.gov/large-docs/16/NCT01647516/SAP_001.pdf